CLINICAL TRIAL: NCT07033962
Title: Comparative Study Between Fractional CO₂ Laser and 40% Urea Assisted Delivery of Topical Fluconazole Microemulsion in the Treatment of Onychomycosis
Brief Title: Fractional CO₂ Laser or 40% Urea With Topical Fluconazole Microemulsion in Onychomycosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shaza Alaa Ezzat Abdel-moneim, doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: onychomycosis treatment
Record Dates: First submitted 2025-05-26; First posted 2025-06-24 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fractional Co2 laser (Experimental): Combination Product:" Fractional CO2 laser" and "topical fluconazole microemulsion"
  Interventions: Combination Product: "Fractional CO2 laser" and "topical fluconazole microemulsion"
- Urea 40% (Experimental): Combination Product: "Urea 40%" and "topical fluconazole microemulsion"
  Interventions: Combination Product: "Urea 40%" and "topical fluconazole microemulsion"

INTERVENTIONS:
Combination Product: "Fractional CO2 laser" and "topical fluconazole microemulsion" — four sessions of fractional CO2 at 3weeks interval with a laser device (multixel, Daeshin enterprise co., LTD. (D.S.E) 105, 271, digital -ro, Guro-gu, Seoul, Koreaa) at a pulse energy of 140 mJ, a density of 150 spots/ cm2 and a depth of 1 cm combined with twice daily topical fluconazole microemulsion.
  Arms: Fractional Co2 laser
Combination Product: "Urea 40%" and "topical fluconazole microemulsion" — urea 40% paste under occlusion once daily over 4 weeks followed by topical fluconazole microemulsion twice daily for 8 weeks.
  Arms: Urea 40%

SUMMARY:
To evaluate the efficacy and safety of topical fluconazole microemulsion enhanced by fractional CO₂ laser versus by 40% urea ablation in treatment of Onychomycosis.

DETAILED DESCRIPTION:
Onychomycosis is a common fungal infection of the nails, caused by dermatophytes, non-dermatophyte molds, and yeasts. The prevalence of onychomycosis is approximately 5.5% of the global population.

Trauma of the nail, aging, nail psoriasis, genetic predisposition and chronic diseases like Diabetes mellitus, immune deficient diseases are considered risk factors for onychomycosis.

Onychomycosis is clinically classified into different types which included:

Subungual onychomycosis which may be proximal (PSO) or distal lateral (DLSO), Endonyx onychomycosis and Total dystrophic onychomycosis (TDO).

Onychomycosis is a contagious disease and will not resolve without treatment leading to deterioration in the quality of life and having the potential to be a source of wider skin infection.

Treatment of onychomycosis includes systemic therapies and topical therapies with or without physical or chemical enhancers.

Topical antifungal medications often fail due to poor nail permeability, while systemic treatments pose risks of hepatotoxicity, drug interactions, and prolonged treatment durations.

Fluconazole is a broad spectrum azole antifungal. It inhibits lanosterol-14-α-demethylase, an enzyme important for the synthesis of ergosterol, a component of fungal cell walls. Compared with other azole derivatives (e.g. ketoconazole, itraconazole, miconazole), fluconazole is less lipophilic (log P = 0.5) and has increased antifungal activity, aqueous solubility (8 mg/mL at 37°C) and higher bioavailability, due to the presence of a halogenated phenyl ring and two triazol rings. Despite its efficacy, its limited solubility and poor nail penetration hinder its topical use. Different topical forms including lipogels, amphiphilogels, hydrogels, emulsions, microemulsions, emulgels, microemulsion gels and liposomal gels have been investigated as vehicles for topical delivery of fluconazole. The topical fluconazole microemulsion-based emulgel has been found to enhance solubility, release, and adherence to the nail.

Fractional CO₂ laser is considered a physical enhancer that creates micro-channels in the nail plate, allowing deeper drug penetration. In addition, it has a direct killing effect of the fungus through photothermal damage. Furthermore, the fractional CO2 laser may contribute to inhibiting fungal growth by causing vaporization and exfoliation of the local tissue around the affected nail.

Similarly, 40% urea acts as a chemical enhancer through its keratolytic agent causing softening and thinning of the nail plate to facilitate drug permeation.

Several studies reported the efficacy of fractional CO2 laser and 40% urea in combination with several topical antifungal treatments as bifonazole and tioconazole in the treatment of onychomycosis. However, no studies have investigated or compared their efficacy in combination with topical fluconazole microemulsion yet.

ELIGIBILITY:
Inclusion Criteria:

* Clinically and mycologically confirmed onychomycosis
* No topical antifungal use in the past 1 month
* No systemic antifungal use in the past 3 months

Exclusion Criteria:

* pregnancy or lactation
* Nail disorders such as psoriasis, eczema, lichen planus
* patients have a known allergy to any of the study treatments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
comparison effect of fractioal co2 laser and 40% urea assisted delivery of topical fluconazole microemulsion in onychomycosis | one month after end of treatment
  Onychomycosis Severity Index (OSI) score will be assessed for each patient Points were given based on :
  1. The percentage of nail involvement (0-5points) 0% 0 point 1-10% 1 point 11-25% 2 points 26-50% 3 points 51-75% 4 points 76-100% 5 points
  2. Proximity of disease to matrix (1-5 points) <25% 1 point, 25-50% 2 points ,50-75% 3 points, >75% 4 point, Matrix involvement 5 points
  3. Dermatophytoma or subungual hyperkeratosis > 2 mm. Present 10 points, Absent 0 points The score will be calculated by this equation: [Score for percentage of involvement * Score for the proximity of disease to the matrix + Score for dermatophytoma or subungual hyperkeratosis > 2 mm] Then the onychomycosis is classified as mild (1-5 points), moderate (6-15 points) or severe (16-35 points), zero indicates cured